CLINICAL TRIAL: NCT05547360
Title: Analysis of Metabolomics of Blood Degradation/Digestion Using in Vitro Digestion Model to Identify Potential Biomarkers of Gastrointestinal Bleeding
Brief Title: Analysis of Blood Metabolomics to Identify Potential Biomarkers of Gastrointestinal Bleeding
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Jung Eun Kim, Assistant professor, National University of Singapore
Other Study IDs: S18
Record Dates: First submitted 2022-09-13; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: GastroIntestinal Bleeding
Keywords: in vitro digestion; Metabolomics; gastrointestinal tract
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite advances in gastrointestinal endoscopy and pharmaceuticals, gastrointestinal bleeding is still a significant emergency disease with a high mortality rate of 1.9-5 per 100 people due to excessive bleeding and shock.

There are several indicators using pulse rate, blood pressure, hemoglobin, etc. to select patients who require endoscopic intervention, or hospitalization, but these are inaccurate and with a high false-positive rate and low specificity at 35-40%.

Therefore, tests with high diagnostic accuracy for gastrointestinal bleeding patients are required and findings specific biomarkers for gastrointestinal bleeding are of great importance.

DETAILED DESCRIPTION:
Recently, with the development of metabolomics, efforts are being made to improve the diagnosis and treatment of diseases through metabolomics analysis, but there are no studies related to gastrointestinal bleeding. If the degradation/metabolism process of blood that accumulates in the gastrointestinal tract is well studied and understood, there is a possibility of finding specific biomarkers for gastrointestinal bleeding.

Thus, this study aims to analysis of metabolomics of blood degradation/digestion using in vitro digestion model to identify potential biomarkers of gastrointestinal bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants, aged between 21 and 55 years old.
2. A body mass index (BMI) between 18.5 and 29.9 kilograms per meter square.
3. English-literate and able to give informed consent in English.

Exclusion Criteria:

1. Smokers.
2. Clinically significant allergic, renal, cardiac, bronchopulmonary, vascular, gastrointestinal, neurological, metabolic or immunodeficiency disorders, cancer, hepatitis, or cirrhosis.
3. Had surgery of the gastrointestinal tract or any other medical condition considered likely to affect the gastrointestinal absorption.
4. Use of oral iron supplement within the past 30 days.
5. Consumes more than 2 alcoholic drinks per day i.e. one drink is defined as either 150ml of wine, 340ml of beer/cider or 45ml of distilled spirit.
6. Significant change in weight (≥ 3 kg body weight) in the past 3 months.
7. Significant exercise pattern over the past 3 months defined as high-intensity exercise of more than 3 hours per week.
8. Poor peripheral venous access based on past experiences with blood draw

Ages: 21 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: Study population are in general good health and not oral consuming iron supplement within the past 30 days.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
blood metabolites | through study completion, an average of 5 months
  screening of blood metabolites in digested blood (qualitative measure, untargeted analysis, using LC-qtof-MS and GC-MS)

CONTACTS AND LOCATIONS:
Overall Officials: Jung Eun Kim, Ph.D, Principal Investigator — National University of Singapore (Food Science and Technology)
Locations (1):
- National University of Singapore, Singapore, Singapore